CLINICAL TRIAL: NCT06756113
Title: Digital Dyadic Empowerment Program (DDEP) on Lifestyle Modification for Chronic Kidney Disease Management: A Randomized Controlled Trial
Brief Title: Digital Dyadic Empowerment Program on Lifestyle Modification for Chronic Kidney Disease Management
Acronym: DDEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Principal Investigator, Miaofen Yen, Professor, Department of Nursing, College of Medicine, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NHRI-EX114-11106PI
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Diseases
Keywords: digital health; dyadic empowerment; healthy lifestyle
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Dyadic Empowerment + Usual Care (Experimental): The intervention group (Digital Dyadic Empowerment + Usual Care) will receive usual care and utilize LINE, a prominent instant messaging App in Taiwan, to assist in lifestyle modification at home along with support from the significant other.
  Interventions: Behavioral: Digital Dyadic Empowerment; Behavioral: Usual Care
- Usual Care (Active Comparator): The control group will receive usual care only.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Digital Dyadic Empowerment — The Digital Dyadic Empowerment Intervention utilizes LINE, a prominent instant messaging App in Taiwan, integrated with an extended application to deliver comprehensive lifestyle modification support to Chronic Kidney Disease (CKD) dyads. Key features of this intervention include:
  1. Access to CKD Health Education Information;
  2. Supportive Information for Significant Others;
  3. Physiological Values Logging for Self-Monitoring;
  4. Reminders for Clinical Appointments and Daily Self-Management Tasks;
  5. Kidney Health Diary for Lifestyle Modification Progress Tracking;
  6. Frequently Asked Questions (FAQs) and Consultation with Healthcare Providers.
  This intervention aims to enhance the overall well-being of CKD dyads by promoting education, self-monitoring, adherence to appointments, and efficient communication with healthcare providers.
  Other Names: LINE Official Account - Kidney Lifestyle
  Arms: Digital Dyadic Empowerment + Usual Care
Behavioral: Usual Care — All patients in this study received regular nephrology care at National Cheng Kung University Hospital. Nephrologists conducted routine examinations and provided diagnoses based on test results. The patient's condition (e.g., changes in kidney function), treatment plan, prognosis, and risks were explained to both the patient and family members. The treatment plan included medication, monitoring blood pressure, dietary and exercise at home, and consultations with the Health Education Center for kidney care or nutrition advice.

SUMMARY:
The goal of this clinical trial is to find out if the Digital Dyadic Empowerment Program (DDEP) can help people with chronic kidney disease (CKD) and their care partners make healthy lifestyle changes. The main questions this study will answer are:

* Does DDEP help protect kidney function?
* Does DDEP support healthier daily habits?

Researchers will compare two groups:

* One group will receive the DDEP and get usual medical care.
* The other group will get usual medical care only.

Participants will:

* Receive usual care with or without DDEP for six months.
* Visit the clinic at the start and end of the study for health checks and tests.
* Practice healthy habits at home with or without help from DDEP.

This study aims to show if adding DDEP to regular care can make it easier for people with CKD and their care partners to live healthier lives.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) aims to evaluate the long-term effects of the Digital Dyadic Empowerment Program (DDEP) in comparison to routine care for people with chronic kidney disease (CKD) and their significant others. The study will assess whether the DDEP can improve health outcomes such as kidney function, health-promoting lifestyle behaviors, and the quality of relationships between significant others over a six-month period. The trial will follow the Consolidated Standards of Reporting Trials (CONSORT) 2010 and CONSORT-EHEALTH guidelines to ensure rigorous reporting and transparency.

Baseline assessments will occur in a private clinic room and will include demographic information, disease-related characteristics, and self-reported measures. Participants in both groups will also complete the Trans-Theoretical Model (TTM) staging inventory to evaluate their readiness for lifestyle changes. Dyads assigned to the intervention group will receive DDEP setup instructions and training on platform use during the baseline visit. Throughout the study, dyads will be encouraged to utilize the platform for self-management tasks at home, including diet tracking, exercise planning, and monitoring blood pressure.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a diagnosis of Chronic Kidney Disease for at least six months;
2. The patient can identify a helpful significant other, and both parties are willing to participate;
3. The patient can communicate in Mandarin or Taiwanese.

Exclusion Criteria:

1. The significant other is a healthcare provider;
2. The patient or the significant other has a mental illness diagnosis;
3. The patient is currently receiving renal replacement therapies;
4. Neither the patient nor the significant other uses a smartphone or the LINE messaging app.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-10-08 (Actual); Study Completion 2025-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miaofen Yen, PhD, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The "Enrollment" number (i.e., 208) in the Study Design Section reflects the total number of *participants* enrolled. After enrollment, 52 dyads (i.e., 52 patients and their 52 significant others) were randomly allocated to each group.
Groups:
- Intervention Group (Digital Dyadic Empowerment + Usual Care): The intervention group (Digital Dyadic Empowerment + Usual Care) will use a platform based on LINE, a prominent instant messaging App in Taiwan. The platform is named "Kidney Lifestyle," consisted of a LINE Official Account (OA) and an extended App.
  The primary objective of Digital Dyadic Empowerment is to encourage CKD dyads (patients and their significant others [SOs]) in modifying health-related lifestyles through the platform and instant messaging support. The main features include:
  1. Health Education Information: Providing basic CKD management knowledge via interactive messages.
  2. Kidney Support Teammate: Offering supportive resources for caregivers (significant others).
  3. Record Values: Allowing users to track physiological measurements at home through the extended App.
  4. Reminders Settings: Automatically sending messages to remind users of outpatient visits and daily self-management tasks.
  5. Kidney Health Mission: Facilitating daily recording of diet, medication intake, and physical activity through the extended App.
  6. Inquiry & Consultation: Providing common CKD-related Q&A and consultation channels through interactive messages.
  The use of the platform is not restricted by time or location, allowing CKD dyads to engage flexibly based on their needs or healthcare providers' instructions. Specifically, users are encouraged to engage daily with two main features, "Record Values" and "Kidney Health Mission," to document their lifestyle modification progress.
- Control Group (Usual Care Only): All study participants received regular checkups and treatments at the nephrology clinics of National Cheng Kung University Hospital. Nephrologists diagnosed and explained disease progression, treatment plans, prognosis, and risks based on clinical assessments. Care plans included medication adherence, home blood pressure monitoring, dietary adjustments, and regular physical activity. Participants also received nephrology nursing or nutritional counseling through the hospital's Health Education Center.
Period: Overall Study
Arm/Group | Intervention Group (Digital Dyadic Empowerment + Usual Care) | Control Group (Usual Care Only)
Started | 104 (After enrollment, 52 dyads (i.e., 52 patients and their 52 significant others) were randomly allocated to each group.) | 104 (After enrollment, 52 dyads (i.e., 52 patients and their 52 significant others) were randomly allocated to each group.)
Completed | 101 | 87
Not Completed | 3 | 17
Not completed — Lost to Follow-up | 3 | 17

BASELINE CHARACTERISTICS:
Population: For each group, there are 52 dyads (i.e., 52 patients and their 52 significant others, totalling 104 participants) for baseline assessment. The overall number of baseline participants is therefore 208 (104*2).
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group (Digital Dyadic Empowerment + Usual Care) | Control Group (Usual Care Only) | Total
Number analyzed (Participants) | 104 | 104 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All 208 participants completed the baseline measure of Age. However, averaging the age of each dyad is not of great interest to our study and could be misleading as the role of the significant other (e.g., the patient's spouse, child, or grandchild) is not taken into account. Therefore, we report the distribution of age for patient and significant other separately.
  years
    Patient: number analyzed (Participants) | 52 | 52 | 104
    Patient | 66.23 (15.19) | 69.81 (12.40) | 68.02 (13.92)
    Significant other: number analyzed (Participants) | 52 | 52 | 104
    Significant other | 57.63 (12.05) | 59.35 (13.22) | 58.49 (12.62)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All 208 participants completed the baseline measure of Sex. However, the count of sex for all participants together is not of great interest to our study and could be misleading as the role of the significant other (e.g., the patient's spouse, child, or grandchild) is not taken into account. Therefore, we report the count of sex for patient and significant other separately.
  Participants
    Patient: number analyzed (Participants) | 52 | 52 | 104
    Patient: Female | 25 | 26 | 51
    Patient: Male | 27 | 26 | 53
    Significant other: number analyzed (Participants) | 52 | 52 | 104
    Significant other: Female | 36 | 31 | 67
    Significant other: Male | 16 | 21 | 37
eGFR [Mean (Standard Deviation); unit: mL/min/1.73m^2] — Estimated Glomerular Filtration Rate (eGFR) by the IDMS-MDRD Equation Population: This measure includes patient only. All 104 patients had baseline eGFR data available. One physiologically implausible value (195.82) from a patient in the intervention group was excluded, leaving 103 datapoints for this measure.
  mL/min/1.73m^2
    number analyzed (Participants) | 51 | 52 | 103
    (all) | 50.69 (23.39) | 46.99 (27.24) | 48.82 (25.35)
CKD Stage [Count of Participants; unit: Participants] — A patient's stage of chronic kidney disease (CKD) based on eGFR. Criteria: Stage 1 (eGFR 90 or above), Stage 2 (eGFR 60-89), Stage 3a (eGFR 45-59), Stage 3b (eGFR 30-44), Stage 4 (eGFR 15-29), Stage 5 (eGFR less than 15). Higher stages (Stage 3b, Stage 4, and Stage 5) represent more advanced and severe progression of chronic kidney disease, with Stage 5 being the most advanced stage. Population: This measure includes patient only. All 104 patients had baseline CKD Stage data available.
  Participants
    number analyzed (Participants) | 52 | 52 | 104
    Stage 1 | 5 | 5 | 10
    Stage 2 | 11 | 8 | 19
    Stage 3a | 11 | 14 | 25
    Stage 3b | 16 | 10 | 26
    Stage 4 | 6 | 8 | 14
    Stage 5 | 3 | 7 | 10
TTM Stage [Count of Participants; unit: Participants] — The TTM stages of change in lifestyle modification were assessed using five statements based on the Transtheoretical Model (TTM). Patients self-assessed their motivation for lifestyle modification, identifying as being in the "precontemplation," "contemplation," "preparation," "action," or "maintenance" stage. Population: This measure includes patient only. All 104 patients had baseline TTM Stage data available.
  Participants
    number analyzed (Participants) | 52 | 52 | 104
    Precontemplation | 1 | 2 | 3
    Contemplation | 2 | 1 | 3
    Preparation | 7 | 1 | 8
    Action | 7 | 13 | 20
    Maintenance | 35 | 35 | 70
Health Promoting Lifestyle [Mean (Standard Deviation); unit: units on a scale] — Patients' lifestyles were assessed using the Health Promoting Lifestyle Profile-II Chinese Revised (HPLP-IICR), a validated scale with 30 items rated on a 4-point Likert scale. The total score ranges from 30 to 120, with higher scores indicating better health-promoting lifestyle. Population: This measure includes patient only. All 104 patients had baseline HPLP-IICR data available.
  units on a scale
    number analyzed (Participants) | 52 | 52 | 104
    (all) | 84.58 (16.74) | 87.23 (15.27) | 85.90 (16.00)
Dyadic Adjustment [Mean (Standard Deviation); unit: units on a scale] — The quality of the relationship between the patient and their significant other was assessed using the 7-item Dyadic Adjustment Scale (DAS-7). The first six items are rated on a 6-point scale, while the seventh item is rated on a 7-point scale, with total scores ranging from 0 to 36. Higher scores indicate better relationship quality. Population: All 208 participants completed the baseline measure of DAS-7. We report the score distribution for patient and significant other separately.
  units on a scale
    Patient: number analyzed (Participants) | 52 | 52 | 104
    Patient | 23.40 (7.08) | 25.71 (7.30) | 24.56 (7.25)
    Significant other: number analyzed (Participants) | 52 | 52 | 104
    Significant other | 21.96 (6.64) | 23.83 (7.46) | 22.89 (7.09)
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in eGFR at 6 Months (Patient-specific)
Description: For each patient, change from Baseline (Followup score - Baseline score) in the estimated Glomerular Filtration Rate (eGFR) by the Isotope Dilution Mass Spectrometry - Modification of Diet in Renal Disease (IDMS-MDRD) Equation at 6 months was obtained through the patient's biochemical test reports. Higher eGFR numbers generally indicate better kidney functions.
Time Frame: Before initial intervention and 6 months after initial intervention
Population: The test of eGFR was conducted only on patient participants. For follow-up, 50 patients from the intervention and 43 patients from the control group completed the eGFR measure.
Measure: Mean (Standard Error); unit: mL/min/1.73m^2
Arm/Group | Intervention Group (Digital Dyadic Empowerment + Usual Care) | Control Group (Usual Care Only)
Number analyzed (Participants) | 50 | 43
mL/min/1.73m^2 | -2.35 (1.31) | -4.24 (1.17)

2. Secondary Outcome: Change From Baseline in CKD Stage at 6 Months (Patient-specific)
Description: For each patient, change from Baseline in CKD stage at 6 months was obtained by comparing the CKD stage at baseline and at follow-up, converted into the following three categories: (1) recover (e.g., from Stage 3a [at baseline] to Stage 2 [at follow-up]); (2) stable (e.g., remaining Stage 3a at both baseline and follow-up); and (3) progress (e.g., from Stage 3a [at baseline] to Stage 3b [at follow-up]).
Time Frame: Before initial intervention and 6 months after initial intervention
Population: The test of CKD Stage was conducted only on patient participants. For follow-up, 50 patients from the intervention and 43 patients from the control group completed the CKD Stage measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group (Digital Dyadic Empowerment + Usual Care) | Control Group (Usual Care Only)
Number analyzed (Participants) | 50 | 43
Participants
  Recover | 6 | 1
  Stable | 37 | 31
  Progress | 7 | 11

3. Secondary Outcome: Change From Baseline in TTM Stage at 6 Months (Patient-specific)
Description: For each patient, change from Baseline in TTM stage at 6 months was obtained by comparing the TTM stage of change at baseline and at follow-up, converted into the following three categories: (1) regress (e.g., from Preparation [at baseline] to Contemplation [at follow-up]); (2) maintain (e.g., remaining Action at both baseline and follow-up); and (3) advance (e.g., from Action [at baseline] to Maintenance [at follow-up]).
Time Frame: Before initial intervention and 6 months after initial intervention
Population: The test of TTM Stage was conducted only on patient participants. For follow-up, 51 patients from the intervention and 44 patients from the control group completed the TTM Stage measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group (Digital Dyadic Empowerment + Usual Care) | Control Group (Usual Care Only)
Number analyzed (Participants) | 51 | 44
Participants
  Regress | 8 | 5
  Maintain | 33 | 33
  Advance | 10 | 6

4. Secondary Outcome: Change From Baseline in Health Promoting Lifestyle at 6 Months (Patient-specific)
Description: For each patient, change from Baseline (Followup score - Baseline score) in patient's Health Promoting Lifestyle at 6 months was assessed using the Health Promoting Lifestyle Profile-II Chinese version Revised (HPLP-IICR), a validated scale with 30 items rated on a 4-point Likert scale. The total scores range from 30 to 120, with higher scores indicate better health-promoting lifestyle.
Time Frame: Before initial intervention and 6 months after initial intervention
Population: This measure was conducted only on patient participants. For follow-up, 51 patients from the intervention and 44 patients from the control group completed the HPLP-IICR measure.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention Group (Digital Dyadic Empowerment + Usual Care) | Control Group (Usual Care Only)
Number analyzed (Participants) | 51 | 44
units on a scale | -1.59 (1.26) | 1.87 (2.17)

5. Secondary Outcome: Change From Baseline in Dyadic Adjustment at 6 Months
Description: For each participant, change from Baseline (Followup score - Baseline score) in Dyadic Adjustment at 6 months was assessed using the 7-item Dyadic Adjustment Scale (DAS-7). The first six items are rated on a 6-point scale, while the seventh item is rated on a 7-point scale. The total scores range from 0 to 36, with higher scores indicating better relationship quality.
Time Frame: Before initial intervention and 6 months after initial intervention
Population: For follow-up, 102 participants (51 patients + 51 significant others) from the intervention and 88 participants (44 patients and 44 significant others) from the control group completed the DAS-7 measure.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention Group (Digital Dyadic Empowerment + Usual Care) | Control Group (Usual Care Only)
Number analyzed (Participants) | 102 | 88
units on a scale | -0.43 (0.62) | -1.22 (0.64)

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, ranging from 151 to 263 days (mean = 179 days, SD = 19.5).
Description: Adverse events were captured by self-report from patients and significant others during in-person or remote (telephone/LINE) contacts throughout follow-up and recorded by research staff. Analyses include all randomized participants. Self-reported medical visits unrelated to the trial's [digital] intervention were documented during follow-up and were reported as general disorders under the 'other adverse events' category.
Arm/Group | Intervention Group (Digital Dyadic Empowerment + Usual Care) | Control Group (Usual Care Only)
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/104
Other Adverse Events (participants affected / at risk) | 5/104 | 1/104
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group (Digital Dyadic Empowerment + Usual Care) (N=104) | Control Group (Usual Care Only) (N=104)
Self-reported medical visit (unrelated) (General disorders) | 5 | 1 — Participant-initiated reports of physical discomfort requiring medical evaluation/treatment during follow-up; events were judged not related to the digital intervention. Examples: hyponatremia, renal cyst, fracture, syncope, dialysis initiation.

LIMITATIONS AND CAVEATS:
1. Follow-up (6 months) may be too short to detect eGFR changes.
2. As a single-center trial, enrolling only dyads with smartphone/LINE access and an available significant other, generalizability is limited.
3. Usage (any log-in) may not capture behavior-change quality, and some questionnaires may be insensitive/misaligned.
4. Models did not adjust key prognostic factors (e.g., age, baseline CKD stage).
5. Platform issues and RA support needs warrant cautious interpretation of use-outcome links.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT06756113/Prot_SAP_000.pdf